CLINICAL TRIAL: NCT03719378
Title: Traditional Intravenous Versus Oral Fluid Management in Total Knee Arthroplasty
Brief Title: Traditional vs Oral Fluid Management in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Principal Investigator, Colorado Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1060593
Record Dates: First submitted 2017-09-06; First posted 2018-10-25 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Fluid Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Fluid (No Intervention): * NPO Clears and Food after midnight.
  * 2 Liters of lactated ringers administered by anesthesia intraoperatively.
  * Postoperatively - 2 Liters of Crystalloid while in PACU and Inpatient Room for a Total of 4 Liters of Crystalloid within 24 hours. (Patient will receive 500 milliliters while in PACU and 1500 milliliters while in their Inpatient Room, for a total of 2 Liters).
  * Normal diet postoperatively.
- Oral Fluid (Experimental): * Pre Operative Oral Fluids (Patients encouraged to drink a minimum of 60 ounces of clear liquid per day for the 3 days prior to procedure.)
  * NPO Food/Milk: none beginning 8 hours prior to procedure time.
  * Pre Operative Oral Fluids (Patients are asked to drink 10 ounces of clear liquid 4 hours prior to their scheduled procedure time.)
  * Preoperative holding area, IV is started in the patient with Lactated Ringers IV fluid at a rate of 75ml/hr. IV fluids will be stopped and hep-locked in the PACU when the patient is taking PO fluid; the total amount of IV fluids is not to exceed 500ml total.
  * PO fluid protocol: a minimum of 60 ounces of liquid per day for 3 days.
  Interventions: Other: Pre Operative Oral Fluids

INTERVENTIONS:
Other: Pre Operative Oral Fluids — Patients will be self hydrating prior to their total knee replacement.
  Arms: Oral Fluid

SUMMARY:
Purpose: Evidence-based guidelines on optimal perioperative fluid management have not been established in patients undergoing orthopaedic surgery. Recent randomized trials in major abdominal surgery suggest that large amounts of IV fluid may increase morbidity and hospital stay. This study will investigate the effects of two regimens of intraoperative fluid management ("traditional" vs. "oral") with physiologic and patient function as primary outcome measures after surgery.

DETAILED DESCRIPTION:
Evidence-based guidelines on optimal perioperative fluid management have not been established in patients undergoing orthopaedic surgery. Typical intraoperative and post-operative fluid management has been arbitrary without evidence based guidelines established following total joint replacement. The investigators have observed many patients post-operatively with side effects such as fluid overload leading to medical complications requiring either prolonged hospitalization or readmission. Additionally, this overload may lead to wound healing complications secondary to fluid shifts which may be devastating in this patient population. Recent randomized trials in major abdominal surgery suggest that large amounts of IV fluid may increase morbidity and hospital stay. Additionally, this increase fluid may be detrimental in patients with anastomosis leading to failure and/or complications in this patient population. The investigators have defined to specific groups of interest to study in this patient population with regards to fluid management. The first group is the "traditional" IV fluid group where the anesthesiologist gives an unspecific amount of fluid intraoperatively and post-operatively the patient gets a set amount of fluid based on "protocol" on the orthopaedic floor (i.e. 75 cc/hour until good oral intake). This is the protocol utilized by most orthopaedic practices throughout the United States. The second group is defined as patients who are given a specific protocol preoperatively to optimize hydration, followed by limited fluids intraoperatively based on physiologic parameters. This study will investigate the effects of two regimens of intraoperative fluid management ("traditional" vs. "oral") with

ELIGIBILITY:
Inclusion Criteria:

• Patients between the ages of 18-75 years old undergoing a primary total knee arthroplasty for a diagnosis of degenerative osteoarthritis who do not meet the exclusion criteria listed below

Exclusion Criteria:

* Volume-dependent cardiac conditions:
* Aortic stenosis
* Pulmonary valve stenosis
* Subaortic stenosis
* Severe Aortic Insufficiency
* Chronic systolic heart failure
* Eisenmeinger Syndrome
* Severe pulmonary HTN
* Chronic or paroxysmal dysrhythmias
* Pre-operative electrolyte abnormalities
* Abnormalities of the HPA (hypothalamic-pituitary axis)
* Stage 3 Chronic Kidney Disease (or worse)
* Patients taking angiotensin receptor blockers (ARB)
* Patients with uncontrolled diabetes mellitus (patient with A1C of 7+ or on insulin)
* Patients whose BMI is > 35 38 or < 19
* Current use of long acting narcotic medication or 3 or more months of daily short acting narcotic medication
* Patients at risk for electrolyte abnormalities, dehydration or intra-operative hypotension. (patients taking angiotensin receptor blockers, ACE inhibitors (48 hours prior to surgery) and Diuretics)
* Patients with severe, untreated or uncontrolled GERD.
* Patients that cannot receive spinal anesthesia (e.g. patient with back fusions)
* Pre-Operative Anemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marjanovic G, Villain C, Juettner E, zur Hausen A, Hoeppner J, Hopt UT, Drognitz O, Obermaier R. Impact of different crystalloid volume regimes on intestinal anastomotic stability. Ann Surg. 2009 Feb;249(2):181-5. doi: 10.1097/SLA.0b013e31818b73dc. PMID 19212167
- [Background] Marjanovic G, Villain C, Timme S, zur Hausen A, Hoeppner J, Makowiec F, Holzner P, Hopt UT, Obermaier R. Colloid vs. crystalloid infusions in gastrointestinal surgery and their different impact on the healing of intestinal anastomoses. Int J Colorectal Dis. 2010 Apr;25(4):491-8. doi: 10.1007/s00384-009-0854-4. Epub 2009 Nov 27. PMID 19943164
- [Background] Kulemann B, Timme S, Seifert G, Holzner PA, Glatz T, Sick O, Chikhladze S, Bronsert P, Hoeppner J, Werner M, Hopt UT, Marjanovic G. Intraoperative crystalloid overload leads to substantial inflammatory infiltration of intestinal anastomoses-a histomorphological analysis. Surgery. 2013 Sep;154(3):596-603. doi: 10.1016/j.surg.2013.04.010. Epub 2013 Jul 19. PMID 23876362

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Fluid: * Pre Operative Oral Fluids (Patients encouraged to drink a minimum of 60 ounces of clear liquid per day for the 3 days prior to procedure.)
  * NPO Food/Milk: none beginning 8 hours prior to procedure time.
  * Pre Operative Oral Fluids (Patients are asked to drink 10 ounces of clear liquid 4 hours prior to their scheduled procedure time.)
  * Preoperative holding area, IV is started in the patient with Lactated Ringers IV fluid at a rate of 75ml/hr. IV fluids will be stopped and hep-locked in the PACU when the patient is taking PO fluid; the total amount of IV fluids is not to exceed 500ml total.
  * PO fluid protocol: a minimum of 60 ounces of liquid per day for 3 days.
  Pre Operative Oral Fluids: Patients will be self hydrating prior to their total knee replacement.
Period: Overall Study
Arm/Group | Traditional Fluid | Oral Fluid
Started | 75 | 75
Completed | 65 | 65
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Fluid | Oral Fluid | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (7.5) | 60.9 (6.8) | 61 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 31 | 33 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
BMI [Mean (Standard Deviation); unit: kg/m^2 (BMI)] | 28.5 (4.9) | 28.1 (4.2) | 28.3 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Patient Weight will be monitored
Time Frame: Change is patients weight from baseline at pre op to two weeks post op.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 64 | 64
pounds | -1.9 (4.4) | -1.6 (4.4)

2. Secondary Outcome: Knee Range of Motion
Description: Measurements will be done with a standard goniometer (Measurements below are shown as the difference from their pre operative base line measurement to the time points below)
Time Frame: Post Op Day 1, 2 Weeks and 6 Weeks Post Op
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
degrees
  Post Op Day 1 | -30.5 (18.5) | -26.7 (16)
  2 Weeks Post Op | -27.9 (17.5) | -25.5 (16.5)
  6 Weeks Post OP | -7.7 (17) | -4.8 (13.2)

3. Secondary Outcome: Leg Anthropometric (Girth) Measurements
Description: measurements will be performed at 5 & 10 cm suprapatellar, midpatella, and 10 cm infrapatellar with the use of a standard tape measure. measurements below show the difference from their pre operative base line measurement to the timepoints below.
Time Frame: Post op Day 1, 2 weeks and 6 weeks Post Op
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
inches
  (10 cm suprapatellar) Post Op day 1 | 2.5 (3.0) | 2.1 (3.1)
  (10 cm suprapatellar) 2 weeks post op | 0.9 (3.0) | 1.6 (4.0)
  (10 cm suprapatellar) 6 weeks post op | 0.00 (2.6) | 0.00 (3.3)
  (5 cm suprapatellar) Post Op day 1 | 4.1 (2.4) | 4.0 (2.6)
  (5 cm suprapatellar) 2 weeks post op | 2.0 (2.3) | 2.8 (2.6)
  (5 cm suprapatellar) 6 weeks post op | 0.9 (1.9) | 1.0 (2.2)
  (Midpatellar) Post Op day 1 | 4.6 (2.2) | 4.1 (2.6)
  (Midpatellar) 2 weeks post op | 2.2 (2.3) | 3.0 (2.0)
  (Midpatellar) 6 weeks post op | 1.3 (1.6) | 1.3 (2.0)
  (10 cm inferior patella) Post Op day 1 | 2.7 (2.7) | 1.5 (4.6)
  (10 cm inferior patella) 2 weeks post op | 0.8 (2.1) | 0.9 (2.3)
  (10 cm inferior patella) 6 weeks post op | -0.2 (1.3) | 0.1 (1.5)

4. Secondary Outcome: Number of Participants With Requiring Transfusions
Description: Post Operative/Intra Operative Transfusions
Time Frame: intra operative, Post Op Day #1 or #2
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Off Wound Complications Post Operative
Description: incidence of wound infection and wound drainage will be assessed and recorded
Time Frame: Up to 6 weeks Post OP
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Thromboembolic Disease
Description: The incidence of thromboembolic events will be recorded.
Time Frame: Post Opeartive until the 6 week follow up appointment
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants | 1 | 0

7. Secondary Outcome: Quadriceps Strength Measure With a Handheld Dynamometer
Description: The strength testing will be calculated using a handheld dynamometer
Time Frame: Post Op day 1, 2 Week and 6 Week Post OP
Measure: Mean (Standard Deviation); unit: KG
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
KG
  Change from Preop to Post Op Day1 | -10.4 (7.6) | -11.2 (7.1)
  Change from Preop to 2 weeks post op | -9.0 (6.5) | -9.6 (7.2)
  Change from Preop to 6 weeks post op | -3.2 (5.8) | -3.8 (6.5)

8. Secondary Outcome: Time up and GO
Description: timed up and go (TUG)
Time Frame: preoperative appointment and once again at their 2 and 6 weeks postoperatively
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Seconds
  Change from Preop to 2 weeks Post op | 4.4 (4.8) | 3.3 (3.7)
  Change from Preop to 6 weeks Post op | -4.7 (3.5) | -4.0 (3.9)

9. Secondary Outcome: 30 Second STS Test
Description: 30 second sit-to-stand tests
Time Frame: preoperative appointment and once again at their 2 and 6 weeks postoperatively
Measure: Mean (Standard Deviation); unit: sit-to-stand events
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
sit-to-stand events
  Change from Preop to 2 weeks Post op | -5.3 (4.0) | -4.4 (4.6)
  Change from Preop to 6 weeks Post op | -0.4 (4.1) | 0.3 (3.0)

10. Secondary Outcome: Length of the Hospitalization
Description: Length of time the patient is Hospitalized after their total knee replacement.
Time Frame: Daily up to 2 days while hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants
  1 Day | 56 | 63
  2 Days | 9 | 2

11. Secondary Outcome: Number of Patients Re-admitted Post TKA
Description: Number of patients re-admitted post TKA
Time Frame: up to 6 weeks post op
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants | 1 | 0

12. Secondary Outcome: Postoperative Pain Assessment Using Visual Analog Scale
Description: Pain will be assessed using a pain Visual Analog scale(VAS), the scale is from 1 to 10, the higher the score the worse the pain.
Time Frame: Every 4 hours, averaged daily, reported at Post op day 1 and 2 (while in the hospital), weeks 1, 2, 3, and 4 (3 times a day)
Population: Some of the patients did not complete their pain log for the study, which is why the numbers are different below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
units on a scale
  Average Post Op Day 1 | 2.6 (1.4) | 2.3 (1.4)
  Average Post Op Day 2: number analyzed (Participants) | 14 | 11
  Average Post Op Day 2 | 4.4 (1.5) | 4.5 (1.6)
  Average Week 1: number analyzed (Participants) | 57 | 60
  Average Week 1 | 4.3 (1.6) | 4.1 (1.6)
  Average Week 2: number analyzed (Participants) | 57 | 58
  Average Week 2 | 3.6 (1.8) | 3.4 (1.5)
  Average Week 3: number analyzed (Participants) | 50 | 53
  Average Week 3 | 3.0 (1.7) | 3.2 (1.7)
  Average Week 4: number analyzed (Participants) | 48 | 48
  Average Week 4 | 2.7 (1.6) | 2.6 (1.4)

13. Secondary Outcome: PONV (Post-operative Nausea and Vomiting)
Description: patients will be asked about Nausea: None, Mild, Moderate or Severe
Time Frame: Daily up to 2 days while hospitalized
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants
  None | 51 | 46
  Mild | 9 | 12
  Moderat | 3 | 3
  Severe | 2 | 4

14. Secondary Outcome: Veterans Rand -12
Description: Patient Reported Outcomes- Veterans Rand(VR-12), there is an algorithm to calculate this score, not a specific range. The higher the number the more positive the output. The score has two components a mental score (MCS) and Physical Score (PCS). Higher values represent a better outcome.
  MCS Scale 35.089613 to 46.341715 PCS Scale 14.957554 to 63.235672
Time Frame: 2 week and 6 week follow up appointments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
score on a scale
  Change from Preop - 2 Weeks Post Op Mental Score | -4.7 (12.2) | -1.2 (10.4)
  Change from Preop - 2 Weeks PostOp Physical Score | -8.3 (10) | -4.5 (11.2)
  Change from Pre op - 6 Weeks Post Op Mental Score | -2.5 (11.5) | -3.2 (11.4)
  Change from Preop - 6 Weeks PostOp Physical Score | -0.5 (10.6) | 2.2 (12.2)

15. Secondary Outcome: Patient Reported Outcomes - Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: Knee injury and Osteoarthritis Outcome Score (KOOS), the scale is 0 to 100, 100 being the best score possible.
Time Frame: pre-operatively as well as at their 2 week and 6 week follow up appointments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
score on a scale
  Change is score from pre op to 2 weeks | -1.6 (16.2) | 3.1 (13.8)
  Change is score from pre op to 6 weeks | 9.4 (14.5) | 12.3 (14.1)

16. Secondary Outcome: Patient Reported Outcomes - Knee Society Score(KSS)
Description: Knee Society Score(KSS), the total scores range from 0 - 200, 200 being the best.
Time Frame: pre-operatively as well as at their 2 week and 6 week follow up appointments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
score on a scale
  Change from Preop to 2 weeks Post op | -14.6 (39.9) | -0.2 (36.2)
  Change from pre op to 6 weeks | 31.9 (36.3) | 40.5 (35.4)

17. Secondary Outcome: Total IV Fluids Received
Description: Total amount of IV fluids that the patients received while in the hospital
Time Frame: Duration of IV intervention, up to 2 days
Measure: Median (Inter-Quartile Range); unit: ML
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
ML | 3895 [1500 to 5322] | 350 [177 to 1466]

18. Secondary Outcome: Bioimpedence
Description: body composition before and after surgery to measure swelling. Lower numbers represent more swelling.
Time Frame: pre-op visit, Post Op Day #1 as well as their 2 week and 6 week visit
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
ohms
  Change from Preop to Post Op Day1 | -17.8 (30.3) | 4.2 (29.7)
  Change from Preop to 2 weeks post op | -41.4 (34.2) | -38.5 (45.7)
  Change from Preop to 6 weeks post op | -30.9 (25.6) | -31.0 (31.4)

19. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: episodes such as symptomatic hypotension (light-headedness, syncope), emesis, the need the IV fluid boluses, and other hospital and post-discharge events will be recorded
Time Frame: While in hospital until the 6 week follow up appointment
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants | 3 | 2

20. Other Pre Specified Outcome: Blood Pressure
Description: Blood Pressure (Diastolic/ Systolic)
Time Frame: Daily up to 2 days while hospitalized
Measure: Mean (Standard Deviation); unit: Change in mmHg
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Change in mmHg
  Change in mmHg Pre Op to Recovery Room (Systolic) | 21.5 (15.9) | 26.0 (16.7)
  Change in mmHg Pre Op to Recovery Room (Diastolic) | 18.4 (12.2) | 17.2 (11.9)
  Change in mmHg Pre Op to Arrival on 4th floor (Systolic) | 10.6 (12.8) | 19.4 (13.5)
  Change in mmHg Pre Op to Arrival on 4th floor (Diastolic) | 10.5 (10.3) | 9.3 (10.8)
  Change in mmHg Pre Op to 08:00 on floor (Systolic) | 17.0 (12.9) | 23.4 (13.3)
  Change in mmHg Pre Op to 08:00 on floor (Diastolic) | 16.5 (9.3) | 16.0 (9.6)
  Change in mmHg Pre Op to 16:00 on floor (Systolic) | 20.9 (14.0) | 25.8 (13.8)
  Change in mmHg Pre Op to 16:00 on floor (Diastolic) | 16.3 (11.2) | 18.7 (11.8)
  Change in mmHg Pre Op to 24:00 on floor (Systolic) | 12.5 (14.7) | 12.5 (12.9)
  Change in mmHg Pre Op to 24:00 on floor (Diastolic) | 14.6 (9.9) | 11.1 (10.2)

21. Other Pre Specified Outcome: Total Number of Patients That Received Any Pressor Drugs
Description: total amount of any pressor drugs given intraoperatively (e.g. Ephedrine and Phenylephrine)
Time Frame: Up to Day 1 Post op
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Fluid | Oral Fluid
Number analyzed (Participants) | 65 | 65
Participants
  Yes | 23 | 22
  No | 42 | 43

ADVERSE EVENTS:
Time Frame: 6 Weeks Post Operatively
Arm/Group | Traditional Fluid | Oral Fluid
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Fluid (N=65) | Oral Fluid (N=65)
acute pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient admired to the ER for an acute pulmonary embolism, this is a known risk of having a TKA, and was not related specifically to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03719378/Prot_SAP_000.pdf